CLINICAL TRIAL: NCT04068636
Title: Sentinel Node Localization in Larynx and Pharynx Cancers After Flexible Endoscopy-guided Tracer Injection: a Feasibility Study.
Brief Title: Sentinel Node in Larynx and Pharynx Cancers
Acronym: FLEX-NODE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FLEX-NODE
Record Dates: First submitted 2019-08-08; First posted 2019-08-28 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Head and Neck Cancer; Lymph Node Metastases
MeSH Terms: conditions — Head and Neck Neoplasms; Lymphatic Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Flexible endoscopy guided SNB in larynx and pharynx cancers. (Experimental): Patients with larynx and pharynx cancers will undergo sentinel node biopsy via flexible endoscopy. In this procedure, a radioactive tracer will be injected at 2-4 sites edging the tumor. A SPECT scan will be performed for visualization of the sentinel node(s).
  Interventions: Procedure: Radioactive tracer injection via flexible endoscopy and SPECT scan for visualization of lymph nodes.

INTERVENTIONS:
Procedure: Radioactive tracer injection via flexible endoscopy and SPECT scan for visualization of lymph nodes. — Flexible endoscopy will be performed by one of two experienced head and neck surgeons. Inspection of larynx and pharynx will be performed to determine the extensions of the tumor in all directions. After local anesthesia, 2-4 peritumoral injections of Tc-99m-nanocolloïd will be given. Ten minutes after injection of Tc-99m-nanocolloïd a SPECT scan will be performed.

SUMMARY:
This study explores the feasibility of sentinel lymph node identification in pharynx and larynx cancers using flexible endoscopy-guided tracer injection.

DETAILED DESCRIPTION:
The presence of lymph node metastases has a large impact on prognosis and treatment in head-and neck cancer (HNC) patients and necessitates treatment intensification. However, despite increased spatial resolution of current imaging techniques, around 20% of patients with a pre-operative clinically negative neck will have occult metastases in the neck dissection specimen. It is therefore that, when patients are treated with radiotherapy, the neck is almost always included in the target volume, also when the tumor is clinically staged N0 (elective neck treatment). As a consequence, large tissue volumes must be treated resulting in significant morbidity such as mucositis, dysphagia, xerostomia and on the long term also hypothyroidism and vascular damage.

If the detection of small lymph node metastases can be improved elective neck treatment may be avoided in at least part of the patients resulting in less toxicity and improved quality of life. One promising approach is the sentinel node procedure. Thus far, the sentinel node procedure is not employed in patients with larynx and pharynx cancers that are treated with primary radiotherapy. One reason is that these tumors are not easily accessible for tracer injection and this needs to be done under general anesthesia. However, in the past few years there has been progress with instrumentation via flexible endoscopy. The ENT-department of Radboudumc has developed expertise with endoscopic biopsy taking and even laser surgery of pharynx and larynx cancers.

The purpose of this study is to explore the feasibility of sentinel lymph node identification in pharynx and larynx cancers using flexible endoscopy-guided tracer injection.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged >18 years.
* Mucosal tumor of the oropharynx, hypopharynx or larynx.
* Patients planned to undergo biopsy via flexible endoscopy.
* Patients planned to undergo curative radiotherapy with or without concurrent chemotherapy.
* Patient provided written informed consent.

Exclusion Criteria:

* Patients who underwent previous surgery or radiotherapy to the neck.
* Patients with airway obstruction causing stridor.
* Prior allergic reaction to Tc-99m-nanocolloïd.
* Pregnancy.
* Unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-03-09 (Actual); Primary Completion 2022-01-11 (Actual); Study Completion 2022-01-11 (Actual)

PRIMARY OUTCOMES:
Generation of SPECT-images of sufficient quality for localization of the sentinel node(s) after peritumoral Tc-99m-nanocolloid injection guided by flexible endoscopy. | The data of each patient will be assessed within 6 months.
  All SPECT images will be assessed qualitatively by concerted consensus between a nuclear medicine physician, head and neck surgeons and a radiation oncologist. Aspects that will be evaluated include:
  * Is there sufficient uptake of tracer for identification and localization of lymph nodes?
  * Does tracer uptake in primary tumor interfere with lymph node identification?
  * Is sentinel lymph node localization consistent with what can be expected with normal, undisturbed lymph node drainage and what is known from the literature?

SECONDARY OUTCOMES:
Feasibility of administering at least 2 peritumoral Tc-99m-nanocolloid injections during one procedure of flexible endoscopy. | The data of each patient will be assesses within 6 months.
  The procedure will be documented on video and will be reviewed by the investigational team for accuracy of tracer injections and learning purposes.
Comparison between sentinel nodes identified by SPECT and sentinel nodes identified by routine CT or MRI. | The data of each patient will be assesses within 6 months.
  All SPECT and CT or MR images will be assessed qualitatively by concerted consensus between a nuclear medicine physician, head and neck surgeons and a radiation oncologist. For this outcome measure the following aspect is visually evaluated: can the lymph nodes identified as sentinel nodes by SPECT also be localized on routine diagnostic imaging (CT, MRI, ultrasound)?

CONTACTS AND LOCATIONS:
Overall Officials: Hans Kaanders, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands